CLINICAL TRIAL: NCT06646016
Title: EPIC - A Phase 2, Randomized, Open-label, Multicenter, Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Extracorporeal Photopheresis (ECP) Versus Best Available Therapy (BAT) in Melanoma or Non-Small Cell Lung Cancer (NSCLC) Patients With Immune-related Colitis Induced by Immune Checkpoint Inhibitor Therapy Who Have Inadequate Response to Steroids
Brief Title: EPIC- Extracorporeal Photopheresis (ECP) for Immune-related Colitis
Acronym: EPIC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Withdrawn by Sponsor prior to Enrollment.
Sponsor: Therakos LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNK60052002
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Immune-related Colitis
Keywords: Melanoma; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Methoxsalen; Infliximab; vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UVADEX in conjunction with extracorporeal photopheresis (Experimental): Participants will receive UVADEX, in conjunction with ECP procedure twice weekly for four weeks and then every other week for 8 weeks during the 12-week treatment period according to the treatment schedule.
  Interventions: Drug: Methoxsalen
- Best available therapy (BAT) (Active Comparator): Participants will receive either infliximab or vedolizumab as per the investigator's choice during the 12-week treatment period.
  Interventions: Drug: Infliximab; Drug: Vedolizumab

INTERVENTIONS:
Drug: Methoxsalen — Sterile solution used in conjunction with photopheresis procedure.
  Other Names: UVADEX®, 20 micrograms per milliliter (mcg/mL)
  Arms: UVADEX in conjunction with extracorporeal photopheresis
Drug: Infliximab — Infliximab will be administered intravenously.
  Other Names: REMICADE®; INFLECTRA®; IXIFI®; RENFLEXIS®; AVSOLA®
  Arms: Best available therapy (BAT)
Drug: Vedolizumab — Vedolizumab will be administered intravenously.
  Other Names: ENTYVIO®
  Arms: Best available therapy (BAT)

SUMMARY:
The photoactivating agent UVADEX (methoxsalen) is used in conjunction with extracorporeal photopheresis (ECP) as an immunomodulatory therapy approved for the treatment of cutaneous T-cell lymphoma. ECP involves collecting whole blood from the patient, separating white blood cells (WBCs) via centrifugation, combining them with UVADEX, and then exposing them to ultraviolet A (UVA) light. All blood components, including the treated WBCs, are then returned to the patient.

Immune Checkpoint inhibitor (ICI) therapy is used to treat different types of cancer, and one major side-effect of ICI therapy is immune-related colitis (ir-colitis). The main purpose of the study is to evaluate the efficacy of UVADEX in conjunction with ECP versus best available therapy (BAT) in participants with melanoma or NSCLC that suffer from ir-colitis with inadequate response to steroids.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with unresectable or metastatic melanoma or unresectable, advanced or metastatic NSCLC, who received ICI treatment with agents like anti-programmed death-1 (PD-1), anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4), and had shown a response to the treatment, based on having a complete response, partial response, or stable disease determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Participants diagnosed with ir-colitis of at least Grade 2 severity based on American Society of Clinical Oncology (ASCO) Guidelines (diarrhea with an increase of ≥4 stools more than at baseline) with other causes of diarrhea and colitis ruled out.
* Participants with endoscopy evidence of ir-colitis based on colonoscopy (modified Mayo Endoscopy Subscore of ≥2).
* Participants with inadequate response to corticosteroids, defined as no improvement in ir-colitis after at least 72 hours of corticosteroid treatment, or relapse of ir-colitis during or after corticosteroid tapering.
* Participants who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2.
* Participants who may become pregnant must have a negative serum pregnancy test, agree to use effective birth control methods during the study and for 30 days after the last treatment, and not be breastfeeding.
* Participants whose sexual partner may become pregnant, must use condoms or other effective contraception, and avoid donating blood, semen, or sperm during the study and for 90 days after the last treatment.
* Participants must agree to wear UVA-absorbing, wrap-around sunglasses and cover exposed skin or use a sunblock (sun protection factor [SPF] ≥ 15) for the 24-hour period following treatment with UVADEX, whether exposed to direct or indirect sunlight.

Exclusion Criteria:

* Presence of irAEs and other than ir-colitis, with severity grade > 2 based on ASCO guidelines.
* Treatment of ir-colitis with any systemic therapy other than corticosteroids.
* Concurrent conditions that might require treatment with corticosteroids ≥ 1 milligram per kilogram body weight per day (mg/kg BW/day) prednisone equivalent.
* Concomitant treatment with any chemotherapy or targeted therapy for malignant melanoma, NSCLC, or other cancers.
* Use of any investigational agent within 5 half-lives of the study treatment.
* Contraindications to study interventions or procedures (UVADEX, the ECP procedure, infliximab, or vedolizumab).
* Known allergic reaction to any component of the investigational agents, 8-methoxsalen (UVADEX), infliximab, or vedolizumab.
* Presence of aphakia or history of light-sensitive diseases such as lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porphyria, xeroderma pigmentosum, or albinism.
* Inability to tolerate the fluid shift associated with the ECP procedure.
* Positive test for human immunodeficiency virus (HIV).
* Positive test for tuberculosis (blood test).
* History of prior allogeneic bone marrow or solid organ transplantation.
* Previous or current malignancies within the last 3 years, other than unresectable or metastatic melanoma or unresectable, advanced, or metastatic NSCLC treated with ICI. Exceptions include adequately treated basal or squamous cell skin cancer.

Note: Other Inclusion/Exclusion criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-06 (Estimated); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Remission of ir-colitis at End of Treatment | Week 12 (diarrhea frequency) / Week 13 (colonic mucosal endoscopy score)
  Composite endpoint of remission measured by diarrhea frequency (CTCAE grade 0 or 1 at Week 12) and colonic mucosal endoscopy score (modified Mayo Score 0 or 1 at Week 13).

SECONDARY OUTCOMES:
Total Duration of Remission for ir-colitis Based on the Criteria for Diarrhea | Week 64
  Duration of remission is the time from when diarrhea improves until the time it comes back (if it does).
Proportion of Participants with Complete Resolution of Diarrhea | Week 12
  Complete resolution of diarrhea refers to normal stool frequency.
Proportion of Participants with Complete Resolution of Colonic Endoscopic Changes | Week 13
  Complete resolution of colonic endoscopic changes refers to no signs of inflammation or damage in the colon.
Proportion of Participants with Corticosteroid-free Clinical Remission | Week 12
  Corticosteroid-free clinical remission is assessed based on the absence of diarrhea and daily corticosteroid dose <5 mg prednisolone or equivalent at week 12.
Changes in the Nancy Score | Week 13
  The Nancy histological index comprises 3 histological items defining 5 grades of disease activity: Grade 0 is absence of significant histological disease; Grade 1 is chronic inflammatory infiltrate with no acute inflammatory infiltrate; Grade 2 is mildly active disease; Grade 3 is moderately active disease; and Grade 4 is severely active disease.
Proportion of Participants with Stool Calprotectin Level <150 micrograms per gram (μg/g) | Week 26
Proportion of Participants with Complete Resolution of Other Symptoms of ir-colitis | Week 64
Time to Complete Resolution of ir-colitis Based on Common Terminology Criteria for Adverse Events (CTCAE) Criteria for Colitis | Week 64
Time to Complete Resolution of Other Specified Immune-related Adverse Events (irAEs) (other than ir-colitis) | Week 64
  The other specified irAEs may include pruritis, rash, inflammatory dermatitis, esophagitis, gastritis, hepatitis, pneumonitis, arthritis, myositis, polymyalgia and nephritis.
Time to Complete Discontinuation of Systemic Corticosteroids for at least 1 Week | Week 12
  This is the time taken by a participant to stop using systemic corticosteroids entirely for at least one week.
Progression Free Survival (PFS) for Melanoma and NSCLC | Week 64
  The approximate time from the start of treatment until the first incidence of cancer worsening or participants dying due to any cause.
Overall Survival (OS) | Week 64
  The approximate time from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Therakos LLC
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No